CLINICAL TRIAL: NCT01800747
Title: Clinical Trial for the Assessment of Delayed Antibiotic Treatment in the Non-complicated Acute Respiratory Tract Infections in Pediatric (Study DAP-Pediatrics)
Brief Title: Clinical Trial for the Assessment of Delayed Antibiotic Treatment in Pediatric (DAP-Pediatrics)
Acronym: DAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Asociacion Colaboracion Cochrane Iberoamericana (Other)
Collaborators: Instituto de Salud Carlos III (Other Government); Ministry of Health, Spain (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAP-Pediatrics
Record Dates: First submitted 2013-02-26; First posted 2013-02-28 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Rhinosinusitis; Acute Bronchitis; Acute Otitis Media; Pharyngotonsillitis
Keywords: Delayed antibiotic treatment; Acute respiratory infections; Pediatrics; Satisfaction
MeSH Terms: conditions — Rhinosinusitis; Bronchitis; Otitis Media; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Antibiotic treatment versus delayed antibiotic treatment
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Direct antibiotic treatment (Active Comparator): The doctor gives to parents an antibiotic prescription for their son's respiratory infection which he should start immediately.
  Interventions: Other: Antibiotic prescription strategies
- No antibiotic treatment (No Intervention): The doctor does not give to parents an antibiotic prescription for their son's respiratory infection.
- Delayed antibiotic prescription (Experimental): The doctor gives to parents an antibiotic prescription for their son's respiratory infection with the advice to use it if needed, in case of worsening of symptoms or not improve.
  Interventions: Other: Antibiotic prescription strategies

INTERVENTIONS:
Other: Antibiotic prescription strategies — The patients enrolled will be randomized between three treatment strategies or arms. Patients randomized to delayed treatment arm or direct treatment, doctors can choose the antibiotic that they consider appropriate depending on such local resistance or practice.
  Arms: Delayed antibiotic prescription; Direct antibiotic treatment

SUMMARY:
The general hypothesis is that delayed antibiotic treatment strategy present similar effectiveness, when compared with non-prescription of antibiotics or the prescription of antibiotics, in the non-complicated acute respiratory tract infections in pediatric patients.

DETAILED DESCRIPTION:
The current project (DAP Pediatrics) is a study that explores the optimization of antibiotic prescribing in our country by evaluating the delayed prescription of antibiotics. The proposed trial will take place in the context of a prior similar study we conducted in adults. The study currently underway is the DAP-Adults study (a randomised controlled trial that evaluates several antibiotic prescribing strategies, including de delayed prescription in uncomplicated acute respiratory infections in adults in primary care).

The aim of this study DAP-Pediatrics (randomized, multicenter parallel) to determine the efficacy and safety of delayed prescription of antibiotics compared to direct prescription and non-prescription of antibiotic in uncomplicated acute respiratory infections in pediatric patients. This 3 arms clinical trial will include 450 children and will evaluate the duration and severity of symptoms, antibiotic consumption, parents' satisfaction, the perceived efficacy of antibiotics and the number of visits generated. The project also includes a qualitative study, by means of structured interviews, to assess the perception and attitudes of parents towards the different treatment strategies and carry out a full analysis of economic evaluation.

ELIGIBILITY:
General Inclusion Criteria:

In this study can be enrolled children (2 to 14 ages) with non-complicated acute respiratory tract infections, including pharyngotonsillitis, rhinosinusitis, acute bronchitis and acute media otitis. The doctors include children with these infections if they have reasonable doubts if they should treat with antibiotics.

General Exclusion Criteria:

* Patients not aged between 2 and 14.
* Patients have participated in the DAP-pediatrics previously.
* Patients are severely affected or patients has been felt severely affected for one week (all time).
* Patients with symptoms and signs suggestive of serious illness or severely affected and/or complications (particularly pneumonia, mastoiditis, peritonsillar abscess, peritonsillar cellulitis, intraorbital or intracranial complications).
* Patients at high risk of serious complications due to prior comorbidity. This includes significant heart disease, lung, kidney, liver or neuromuscular, immunosuppression, cystic fibrosis.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-06-07 (Actual)

PRIMARY OUTCOMES:
Duration and severity of symptoms | 30 days
  Coordination Centre performed telephone interviews.

SECONDARY OUTCOMES:
Antibiotic consumption | 30 days
  Self-reported by the patients and checked at the Regional Pharmacy's Units.
Parents satisfaction with treatment | 30 days
  Likert scale.
Parents' belief in the efficacy of antibiotics | 30 days
  Likert scale
Impact of DAP strategy on the reconsultation | 1 year
  Medical history review
The prescription of antibiotics in the previous two years predicts the effect of prescribing strategies in reconsultation. | 1 year
  Medical history review

OTHER OUTCOMES:
Complications of disease | 30 days
  Included by doctors or coordination centre

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Alonso Coello, PhD, Principal Investigator — Asociación Colaboración Cochrane Iberoamericana
Locations (1):
- Asociación Colaboración Cochrane Iberoamericana, Barcelona, Spain

REFERENCES:
- [Derived] Mas-Dalmau G, Perez-Lacasta MJ, Alonso-Coello P, Gorrotxategi-Gorrotxategi P, Arguelles-Prendes E, Espinazo-Ramos O, Valls-Duran T, Gonzalo-Alonso ME, Cortes-Viana MP, Menendez-Bada T, Vazquez-Fernandez ME, Perez-Hernandez AI, Munoz-Ortiz L, Villanueva-Lopez C, Little P, de la Poza-Abad M, Carles-Lavila M; DAP Paediatrics Group. A trial-based cost-effectiveness analysis of antibiotic prescription strategies for non-complicated respiratory tract infections in children. BMC Pediatr. 2023 Oct 2;23(1):497. doi: 10.1186/s12887-023-04235-3. PMID 37784098